CLINICAL TRIAL: NCT02427698
Title: Comparison of the Efficacy Between Cryolipolysis Versus Cryolipolysis Plus Subcision For Treatment of Cellulite: A Prospective Randomized Control Trial
Brief Title: Cyrolipolysis vs Cyrolipolysis and Subcision for Cellulite
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Zeltiq Aesthetics (Industry)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU200346
Record Dates: First submitted 2015-04-13; First posted 2015-04-28 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cyrolipolysis (Active Comparator)
  Interventions: Procedure: cyrolipolysis (CoolSculpting device)
- cryolipolysis plus subcision (Active Comparator)
  Interventions: Procedure: cyrolipolysis (CoolSculpting device); Procedure: subcision

INTERVENTIONS:
Procedure: cyrolipolysis (CoolSculpting device) — Treatment will be a cold exposure for up to 120 minutes using the CoolSculpting device with a commercially available treatment setting.
Procedure: subcision — The skin will be punctured using a subcision needle to cut the septa responsible for the skin depression after cryolipolysis.
  Arms: cryolipolysis plus subcision

SUMMARY:
This is a prospective randomized controlled study comparing the efficacy of cryolipolysis versus a combination of cryolipolysis and surgical subcision for the treatment of cellulite. The treatment sites are both outer thighs. One outer thigh will be randomized to receive one treatment of cryolipolysis, while the contralateral thigh will be assigned to receive the combination cryolipolysis plus surgical subcision. A live rating by a blinded dermatologist will evaluate the treatment and control areas using a cellulite severity scale at week 0 (before treatment) and at the 3-month follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects 18-65 years of age with at least a 5 on the CSS scale on both outer thighs.
2. All subjects must have the affected areas that show the mattress phenomenon spontaneously when standing or while both lying and standing (Stage 2 or 3 of Nurnberger-Muller grading scale of cellulite7).
3. Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator.

Exclusion Criteria:

1. Subjects who are pregnant or lactating.
2. Subjects who are unable to understand the protocol or to give informed consent.
3. Subjects currently under treatment with an antiplatelet or anticoagulant for any medical problem or patients who have coagulation disorder.
4. Subjects who have a known history of cold-induced disease such as cryoglobulinemia, paroxysmal cold hemoglobulinuria, cold urticaria.
5. Subjects who have active skin disease or skin infection in the treatment area.
6. Subjects who are allergic to lidocaine or prilocaine.
7. Subjects who are allergic to both cephalexin (or penicillin) AND levofloxacin (or another quinolone antibiotic).
8. Subjects who have history of abnormal scarring.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Live rating by a blinded dermatologist using cellulite severity scale | Change from Baseline in cellulite severity scale at 3 months
  The cellulite severity scale rates cellulite 1-5 as mild, 6-10 as moderate, and 11-15 as severe.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States